CLINICAL TRIAL: NCT02204111
Title: Patient Directed Intervention Towards a Multidimensional Recommendation Guideline to Improve the Quality of Life for Patients With Soft Tissue Sarcoma Under Palliative Treatment With Trabectedin
Brief Title: Patient Directed Intervention to Improve the Quality of Life for Patients With Soft Tissue Sarcoma
Acronym: YonLife
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: YonLife-2014
Record Dates: First submitted 2014-07-09; First posted 2014-07-30 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Soft Tissue Sarcoma
Keywords: Palliative Treatment; Trabectedin; Patient Reported Outcome
MeSH Terms: conditions — Sarcoma | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Cluster: Care as usual
- Treatment Cluster: Care as usual and patient directed, multidimensional treatment proposals
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Individualized treatment proposals (e.g. pain therapy, physiotherapy, psychological contact) from expert consensus, based on Patient Reported Outcomes
  Groups: Treatment Cluster

SUMMARY:
The primary objective of the study is to compare quality of life (QoL) between patients suffering from soft tissue sarcoma, receiving a multidimensional intervention with those receiving standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or metastatic soft tissue sarcoma
* Treatment with trabectedin in an in-label prescription
* Age at least 18 years (inclusive) at the first visit
* Patients with a life expectancy of at least 6 months
* The informed consent form must be signed before any study specific tests or procedures are done
* Confirmation of the subject's health insurance coverage prior to the first visit
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* ECOG PS >2
* Estimated life expectancy of less than 6 months
* Patients with STS not receiving trabectedin
* Contraindications according to the local SmPC of Yondelis®
* Subject is in custody by order of an authority or a court of law
* Exclusion periods from other studies or simultaneous participation in other clinical studies
* Previous assignment to treatment during this study
* Close affiliation with the investigator (e.g. a close relative) or persons working at the study site
* Subject is an employee of GWT-TUD GmbH or Pharma Mar S.A.
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Soft Tissue Sarcoma under palliative treatment with Trabectedin
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Health related QoL, measured by total score of FACT-G | change to baseline at 9 weeks
  assessed by the patient using standard questionnaire (FACT-G) via tablet-PC

SECONDARY OUTCOMES:
Dimensions of QoL (scales of FACT-G) | baseline, 3, 6, 9, 21, 35 and 61 weeks
  assessed by the patient using standard questionnaire (FACT-G) via tablet-PC
Anxiety and depression (HADS) | baseline, 9, 21, 35 and 61 weeks
  assessed by the patient using standard questionnaire (HADS) via tablet-PC
Satisfaction with care (IN-PATSAT32) | baseline, 9, 21, 35 and 61 weeks
  assessed by the patient using standard questionnaire (IN-PATSAT32) via tablet-PC
Anorexia and cachexia related impact on QoL (FAACT) | baseline, 9, 21, 35 and 61 weeks
  assessed by the patient using standard questionnaire (FAACT) via tablet-PC
Intensity of pain and pain related interference (BPI) | baseline, 9, 21, 35 and 61 weeks
  assessed by the patient using standard questionnaire (BPI) via tablet-PC
Severity of cancer-related symptoms (MDASI) | baseline, 3, 6, 9, 21, 35 and 61 weeks
  assessed by the patient using standard questionnaire (MDASI) via tablet-PC
progression free survival | baseline up to 61 weeks
Overall survival | baseline up to 61 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuler, Dr. med., Principal Investigator — University Hospital Carl Gustav Carus, Dresden
Locations (7):
- Germany (7):
  - University Hospital Carl Gustav Carus, MK I, Dresden, Saxony
  - Charité, Berlin
  - University Hospital Koeln, Cologne
  - Hannover Medical School, Hanover
  - University Medical Centre Mannheim, Mannheim
  - University Hospital Muenster, Münster
  - University Hospital Tuebingen, Tübingen

REFERENCES:
- [Derived] Hentschel L, Richter S, Kopp HG, Kasper B, Kunitz A, Grunwald V, Kessler T, Chemnitz JM, Pelzer U, Schuler U, Freitag J, Schilling A, Hornemann B, Arndt K, Bornhauser M, Schuler MK. Quality of life and added value of a tailored palliative care intervention in patients with soft tissue sarcoma undergoing treatment with trabectedin: a multicentre, cluster-randomised trial within the German Interdisciplinary Sarcoma Group (GISG). BMJ Open. 2020 Aug 27;10(8):e035546. doi: 10.1136/bmjopen-2019-035546. PMID 32859662
- [Derived] Schuler M, Richter S, Ehninger G, Bornhauser M, Hentschel L. A cluster-randomised, controlled proof-of-concept study to explore the feasibility and effect of a patient-directed intervention on quality of life in patients with advanced soft tissue sarcoma. BMJ Open. 2017 Jun 30;7(6):e014614. doi: 10.1136/bmjopen-2016-014614. PMID 28667207